CLINICAL TRIAL: NCT04201379
Title: Nonspecific Neck Patients's Quality of Life and Their Predictors
Brief Title: Determines of Quality of Life in Patients
Status: Completed | Type: Observational
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ayça Aytar TIĞLI, Physical therapist Phd, Baskent University
Other Study IDs: KA19/406
Record Dates: First submitted 2019-11-28; First posted 2019-12-17 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2019-01

CONDITIONS: Chronic Neck Pain
Keywords: chronic; neckpain
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neck pain patients: servical disk hernisi servical spondilosis servical problems
  Interventions: Other: quality of life assesment
- control: healthy people
  Interventions: Other: quality of life assesment

INTERVENTIONS:
Other: quality of life assesment — The sociodemographic and clinical characteristics of the individuals who meet the study criteria will be recorded. Evaluations of the participants will be done only once

SUMMARY:
Pain, muscle spasm, loss of muscle strength and impaired posture adversely affect the daily life activities and quality of life of neck pain patients.However, the quality of life; It is a multifaceted concept that includes not only the age, sex, marital status, educational status and duration of pain, but also the number of children, BMI, depression, sleep quality, pain-related inadequacy and fatigue. Therefore, considering all these; quality of life; The aim of our study was to determine the factors affecting the quality of life in nonspesific neck patients with the effect that the determinants affecting physical, physical role difficulty, pain, general health, vitality, social function, emotional role difficulty and mental health may be different.

DETAILED DESCRIPTION:
The study will include 93 people with a diagnosis neck disease who apply to the physical therapy outpatient clinic. After recorded sociodemographic and clinical characteristics of the individuals, some evaluations will be done only once. The evaluations to be used in the study are as follows: Pain Assesment will be evaluated with McGill Pain Questionnaire, Sleep disorders will be evaluated with Pitsburgh Sleep Quality Index (PSQI), Fatigue level will be assessed by the Fatigue Questionnaire, Beck Depression Inventory (BDI) will be used to determine depression levels. The quality of life of the subjects wiil be evaluate by using the Short Form-36 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1) People 18 years and older

Exclusion Criteria:

1. Hospitalized people
2. Newly Operated People
3. People with psychological diagnosis

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: people with a diagnosis of neck disease living in Ankara and who can answer the study questions
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-04-25 (Actual)

PRIMARY OUTCOMES:
DETERMINING FACTORS AFFECTING THE QUALITY OF LIFE | 27 february 2020
  to reported determining factors affecting their quality of life Short form-SF36 .All questions are scored on a scale from 0 to 100, with 100 representing the highest level of functioning possible. Aggregate scores are compiled as a percentage of the total points possible, using the RAND scoring table (STEP I chart).
  The scores from those questions that address each specific area of functional health status (STEP II chart) are then averaged together, for a final score within each of the 8 dimensions measured. (eg pain, physical functioning etc.)
IS PAIN DETERMINING THE QUALITY OF LIFE | 27 february 2020
  MCMcGill Pain Questionnaire will be used to report pain.The McGill Pain Questionnaire (MPQ) is a three-part pain assessment tool that measures several dimensions of the patient's pain experience. The first part consists of an anatomic drawing of the human form on which the patient marks where his or her pain is located. The second part of the MPQ is a VDS that allows the patient to record the intensity level of his or her current pain experience. The third part of the MPQ is a pain verbal descriptor inventory consisting of 72 descriptive adjectives. The patient is asked to review this list of pain descriptors and circle the ones that serve to best describe his or her current pain experience. Each part or dimension of the MPQ is individually scored and a cumulative total score is also recorded.
IS PAIN INTENSITY DETERMINING THE QUALITY OF LIFE | 27 february 2020
  Visual Analog Score for pain, Physicians Global Assessment to measure quality of life.The pain VAS is a continuous scale comprised of a horizontal (HVAS) or vertical (VVAS) line, usually 10 centimeters (100 mm) in length, anchored by 2 verbal descriptors, one for each symptom extreme .r pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale])
IS SLEEP QUALİTY DETERMINING THE QUALITY OF LIFE | 27 february 2020
  te report the effect of sleep quality Pitsburgh Sleep Quality Index will be used. The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep in the older adult. It differentiates "poor" from "good" sleep by measuring seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. The client self rates each of these seven areas of sleep. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale. A global sum of "5"or greater indicates a "poor" sleeper
IS FATIGUE DETERMINING THE QUALITY OF LIFE | 27 february 2020
  Fatigue Questionnaire will be used to report fatigue.Scoring using a bimodal response system or a Likert score with weights assigned to each response choice. Likert or bimodal rating scales with 4 response options. For the Likert Scale: better than usual = 0, no more than usual = 1, worse than usual = 2, much worse than usual = 3. For the bimodal scale: better than usual = 0, no more than usual = 0, worse than usual = 1, much worse than usual = 1. Sum all items for a total score.
IS DEPRESSION DETERMINING THE QUALITY OF LIFE | 27 february 2020
  to report depression levels Beck Depression Inventory (BDI) will be used.Each of the four multiple choice answers is assigned a point value from 0 to 3. At the end of the assessment, you add up the total points from the answers throughout the 21 questions. Hıgh scores ındıcate worse depressıon levels
IS Anxıety DETERMINING THE QUALITY OF LIFE | 27 february 2020
  te report the effect of anxıety State-Trait Anxiety Inventory (STAI) will be used.The higher the score, the higher the level of anxiety.
Is pain disability DETERMINING THE QUALITY OF LIFE | 27 february 2020
  to report disability levels we will be used The Pain Disability Index.High score indicates high disability

CONTACTS AND LOCATIONS:
Locations (1):
- Ayça Aytar, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided